CLINICAL TRIAL: NCT03908905
Title: Prevalence of Sleep Disturbances in Individuals With Chronic Widespread Pain
Brief Title: Sleep Disturbances and Chronic Widespread Pain
Acronym: POSEIDON
Status: Suspended | Type: Observational
Why Stopped: Lack of resources
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00018
Record Dates: First submitted 2019-04-08; First posted 2019-04-09 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Chronic Widespread Pain; Sleep Disturbance
Keywords: Pain; Sleep; Neuropsychology; Fatigue; Activity level; Attention; Executive function; Memory
MeSH Terms: conditions — Chronic Pain; Parasomnias; Pain; Fatigue | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention
  Interventions: Diagnostic Test: Polysomnography

INTERVENTIONS:
Diagnostic Test: Polysomnography — Sleep screening, neurocognitive assessment, activity monitoring questionnaires, blood sample

SUMMARY:
Chronic widespread pain (CWP), defined as long-lasting pain in multiple body regions, has a prevalence of 10-14% in Europe and is associated with other physical symptoms such as fatigue and cognitive problems. Individuals with longstanding pain also have a high prevalence of sleep disturbances, and sleep problems can in itself lead to tiredness, lower neurocognitive function and higher pain ratings. However, studies of comorbid sleep problems for individuals with CWP are a lacking, and the primary aim for the present study is to assess the prevalence of sleep disturbances in individuals with CWP, and to see how this covariates with pain, fatigue, activity level, neurocognitive functioning, and biomarkers. As a secondary aim the study will assess a subgroup of the individuals, that has received multimodal pain management treatment, a second time after 6 months to analyze how the prevalence of sleep disturbances and other associated problems covaries over time.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Widespread Pain

Exclusion Criteria:

* Other untreated and or serious psychiatric or somatic conditions

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All subjects that are referred for an inpatient multidisciplinary analysis of complex chronic pain conditions at a regional pain center at Uppsala University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Polysomnography | 6 months
  Assessment of objective sleep problems

SECONDARY OUTCOMES:
CANTAB | 6 months
  Neurocognitive screening
Actigraph | 6 months
  Activity level
Biomarkers | 6 months
  92-plex inflammatory panel
Pain level | 6 months
  The Brief Pain Inventory - Short Form, BPI, a 9 item (0-10) self-administered questionnaire, assessing the severity of a patient's pain and the impact of this pain on the patient's daily functioning. Maximum total score possible is 90. Higher the score, greater the degree of disability.
Fatigue | 6 months
  Fatigue severity scale, FSS, a 9 item self-administered questionnaire assessing severity of fatigue and how fatigue interferes with activity. Items are scored on a 7 point scale, minimum total score possible is 9 and maximum 63. Higher the score, greater the severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala university hospital, Uppsala, Uppsala County, Sweden